CLINICAL TRIAL: NCT03770013
Title: Role of Co-administered Dexmedetomidine Or Clonidine With Bupivacaine for Transversus Abdominis Plane Block in Patients Undergoing Elective Caesarean Section: A Randomized, Double-blind Controlled Trial
Brief Title: Dexmedetomidine Versus Clonidine for Transversus Abdominis Plane Block in Patients Undergoing Elective Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/182/18
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain
Keywords: Bupivacaine; Dexmedetomidine; Clonidine; Transversus Abdominis Plane Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexmedetomidine; Clonidine

STUDY DESIGN:
Intervention Model Description: A prospective Randomized Interventional double-blind study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bupivacaine 0.25% and Dexmedetomidine (Active Comparator): bupivacaine 0.25% + Dexmedetomidine 0.5 mcg/kg (a total volume of 40 ml (20 ml each side) was used for the TAP block.)
  Interventions: Drug: bupivacaine; Drug: Dexmedetomidine
- bupivacaine and clonidine (Active Comparator): 20 ml bupivacaine+1ug/kg clonidine bilaterally (a total volume of 40 ml (20 ml each side) was used for the TAP
  Interventions: Drug: bupivacaine; Drug: clonidine
- bupivacaine and placebo (Placebo Comparator): bupivacaine 0.25% + placebo (a total volume of 40 ml (20 ml each side) was used for the TAP
  Interventions: Drug: bupivacaine; Drug: placebo

INTERVENTIONS:
Drug: bupivacaine — bupivacaine 0.25% a total volume of 40 ml (20 ml each side
  Other Names: Active Comparator
Drug: Dexmedetomidine — Dexmedetomidine 0.5 mcg/kg
  Other Names: Active Comparator
  Arms: bupivacaine 0.25% and Dexmedetomidine
Drug: clonidine — 1ug/kg clonidine
  Other Names: Active Comparator
  Arms: bupivacaine and clonidine
Drug: placebo — add placebo 9normal saline)
  Other Names: placebo comparator
  Arms: bupivacaine and placebo

SUMMARY:
Aim to study the efficacy of co-administered Dexmedetomidine Or Clonidine with Bupivacaine and that of bupivacaine 0.25% alone for Transversus Abdominis Plane (TAP) Block for Postoperative Analgesia in Patients Undergoing Elective Caesarean Section.

* Group 1: bupivacaine 0.25% + Dexmedetomidine 0.5 mcg/kg (a total volume of 40 ml (20 ml each side) was used for the TAP block.)
* Group 2: 20 ml bupivacaine+1ug/kg clonidine bilaterally (a total volume of 40 ml (20 ml each side) was used for the TAP
* Group3: bupivacaine 0.25% + placebo (a total volume of 40 ml (20 ml each side) was used for the TAP A prospective Randomized Interventional double-blind study.

DETAILED DESCRIPTION:
Women, following Caesarean delivery, have even more compelling reasons to receive optimal post-operative pain relief, for improved maternal and neonatal well-being. Also, adequate pain relief helps the patient to ambulate early and prevent any thrombotic incidents . Dexmedetomidine, an imidazole compound, is the pharmacologically active dextroisomer of medetomidine that displays specific and selective α 2-adrenoceptor agonist activity and causes sedation, analgesia without any delirium, or respiratory depression. The mechanism of action is unique and differs from those of currently used agents, including clonidine.

ELIGIBILITY:
Inclusion Criteria:

* parturients scheduled to undergo cesarean section under spinal anesthesia

Exclusion Criteria:

* Patients who refused spinal anesthesia
* women with chronic pelvic pain or on chronic morphine use
* history of drug allergy
* coagulation disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients Undergoing Elective Caesarean Section.
Enrollment: 150 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
The time for first rescue analgesia after the TAP block | 24 hours post operative
  calculation the time needed for first rescue analgesia after the TAP block

SECONDARY OUTCOMES:
Total dose of rescue analgesia | 24 hours postoperative
  calculation of Total dose of rescue analgesia required in 24 h post-operatively
Adverse effects | 24 hours postoperative
  Adverse effects like pruritus, nausea and vomiting, hypotension, bradycardia, and sedation.

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided